CLINICAL TRIAL: NCT05786989
Title: Selinexor Combined With R-GemOx as Second-line Treatment in Patients With Diffuse Large B-cell Lymphoma： a Single-arm, Single-centre, Open-label Trial
Brief Title: Selinexor Combined With R-GemOx as Second-line Treatment in Patients With Diffuse Large B-cell Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yao Liu, Chief physician, Chongqing University Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chongqingcancer v3.0_20220908
Record Dates: First submitted 2023-03-02; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Diffuse Large B-Cell Lymphoma, Not Otherwise Specified
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients will receive selinexor PO on days 1, 8, and 15 of a 21 week cycle. R-GemOx will be given at standard dosing every 21 days
  Interventions: Drug: selinexor

INTERVENTIONS:
Drug: selinexor — Given PO
  Other Names: Selective Inhibitor of Nuclear; KPT-330

SUMMARY:
The goal of this interventional study is to evaluate efficiency and safety in prior one-line treated diffuse large B-cell lymphoma. The main questions it aims to answer are:

* Complete remission rate
* Objective remission rate
* Progression-free survival
* tolerance Participants will recevied a minimum of 2 and a maximum of 6 cycles of R-GemOx(rituximab 375 mg/m2 IV on day 1 , Gemcitabine 1000 mg/m2, Oxaliplatin 100 mg/m2 IV on day 2) and 60 mg selinexor on days 1, 8, and 15 of each cycle

DETAILED DESCRIPTION:
After the subject has completed at least 2 courses of treatment with Serenixol and R-GemOx for up to 6 courses, the patients who have reached ≥ partial remission (PR) and meet the conditions of transplantation can receive transplantation according to the institutional standards, and those who are not suitable for transplantation can receive maintenance treatment with Serenixol. In the maintenance treatment, the dose of Serenixol is 60 mg on the first day of the week until the disease progresses In case of intolerable toxicity or if the researcher believes that the patient is no longer suitable for study treatment, re-examine every 3 months in the first year, the second year and every 6 months after the end of transplantation or maintenance treatment; Patients with stable disease (SD) or disease progression (PD) after 2~6 courses of treatment will end the trial, and no survival follow-up will be conducted

ELIGIBILITY:
Inclusion Criteria:

* Have pathologically confirmed CD20 positive de novo DLBCL or DLBCL transformed from previously diagnosed indolent lymphoma (e.g., follicular lymphoma)
* HIV-seropositive
* Age 18-75 years
* ECOG PS≤2
* Positron emission tomography (PET) positive measurable disease with at least one node having the longest diameter (LDi)>1.5cm or one extranodal lesion with LDi>1cm (per the Lugano Criteria 2014) (Documentation to be provided)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 × Upper limit of normal value (ULN), or ≤ 5 in the presence of known lymphoma involving the liver × ULN; Total serum bilirubin ≤ 2 × ULN, or ≤ 5 when Gilbert syndrome or known lymphoma affects the liver × ULN; Creatinine clearance (CrCl) calculated according to Cockcroft Gault formula ≥ 30 mL/min;
* Absolute neutrophil count (ANC)≥1.5×10^9/L,or Platelet count≥75×10^9/L(No platelet were transfused within 14 days before the treatment of the study drug),or Hemoglobin≥80g/L(No red blood cells were transfused within 14 days before the treatment of the study drug)
* Written informed consent in accordance with federal, local, and institutional guidelines
* Patients understanding the characteristics of the disease and voluntarily joins the study program for treatment and follow-up
* No other serious diseases in conflict with this program
* Investigator believe that subjects can benefit

Exclusion Criteria:

* Patients with known central nervous system involvement by lymphoma;
* Patients with a history of autoimmune diseases or syndrome requiring systemic use of steroid, such as hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism and hypothyroidism
* Patients received systemic glucocorticoid (prednisone >20mg/d) or any other immunosuppressive therapy within 7 days before the first administration,excluding nasal spray inhalation or other topical glucocorticoids;
* Uncontrolled heart diseases, including unstable angina pectoris, acute myocardial infarction 6 months before randomization, congestive heart failure (NYHA), cardiac function grade greater than grade III or IV, or left ventricular ejection fraction<50%;
* Patients previously treated with selinexor;
* History of severe allergic reactions (as determined by treating physician) attributed to the drugs being used in the study;
* Patients undergoing organ transplantation;
* Diagnosed as malignant tumor other than lymphoma or receiving treatment,excluding:

  1. Malignant tumors that have received treatment for the purpose of cure and have not developed known active diseases for ≥ 5 years before enrollment
  2. Basal cell carcinoma of the skin (excluding melanoma) with adequate treatment and no signs of disease
  3. Cervical carcinoma in situ with adequate treatment and no signs of disease
* Patients with grade 2 or more neurotoxicity occurred within two weeks before treatment;
* Severe infection;
* Drug abuse, medical psychological or social conditions that may interfere with the subject's participation in the study or the evaluation of the results of the study;
* Any active, serious psychiatric, medical, or other conditions/situations which, in the treating physician's opinion, could compromise the patient's safety

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | UP to 2 years
  Response rates will be estimated as proportions with 95% Wilson confidence intervals

SECONDARY OUTCOMES:
Progression-free survival | From baseline to disease progression or death from any cause, assessed up to 2 years
  PFS will be described with Kaplan-Meier curves and estimated medians with 95% confidence intervals
Objective remission rate | UP to 2 years
  Response rates will be estimated as proportions with 95% Wilson confidence intervals

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
After the paper is published

REFERENCES:
- [Result] Krok-Schoen JL, Fisher JL, Stephens JA, Mims A, Ayyappan S, Woyach JA, Rosko AE. Incidence and survival of hematological cancers among adults ages >/=75 years. Cancer Med. 2018 Jul;7(7):3425-3433. doi: 10.1002/cam4.1461. Epub 2018 Apr 13. PMID 29654631
- [Result] Harris LJ, Patel K, Martin M. Novel Therapies for Relapsed or Refractory Diffuse Large B-Cell Lymphoma. Int J Mol Sci. 2020 Nov 13;21(22):8553. doi: 10.3390/ijms21228553. PMID 33202794
- [Result] Crump M, Neelapu SS, Farooq U, et al. Outcomes in refractory diffuse large B-cell lymphoma: results from the international SCHOLAR-1 study. Blood. 2017;130(16):1800-1808. Blood. 2018 Feb 1;131(5):587-588. doi: 10.1182/blood-2017-11-817775. No abstract available. PMID 29437609
- [Result] Pfreundschuh M, Trumper L, Osterborg A, Pettengell R, Trneny M, Imrie K, Ma D, Gill D, Walewski J, Zinzani PL, Stahel R, Kvaloy S, Shpilberg O, Jaeger U, Hansen M, Lehtinen T, Lopez-Guillermo A, Corrado C, Scheliga A, Milpied N, Mendila M, Rashford M, Kuhnt E, Loeffler M; MabThera International Trial Group. CHOP-like chemotherapy plus rituximab versus CHOP-like chemotherapy alone in young patients with good-prognosis diffuse large-B-cell lymphoma: a randomised controlled trial by the MabThera International Trial (MInT) Group. Lancet Oncol. 2006 May;7(5):379-91. doi: 10.1016/S1470-2045(06)70664-7. PMID 16648042
- [Result] Cunningham D, Hawkes EA, Jack A, Qian W, Smith P, Mouncey P, Pocock C, Ardeshna KM, Radford JA, McMillan A, Davies J, Turner D, Kruger A, Johnson P, Gambell J, Linch D. Rituximab plus cyclophosphamide, doxorubicin, vincristine, and prednisolone in patients with newly diagnosed diffuse large B-cell non-Hodgkin lymphoma: a phase 3 comparison of dose intensification with 14-day versus 21-day cycles. Lancet. 2013 May 25;381(9880):1817-26. doi: 10.1016/S0140-6736(13)60313-X. Epub 2013 Apr 22. PMID 23615461
- [Result] Arboe B, Olsen MH, Gorlov JS, Duun-Henriksen AK, Dalton SO, Johansen C, de Nully Brown P. Treatment intensity and survival in patients with relapsed or refractory diffuse large B-cell lymphoma in Denmark: a real-life population-based study. Clin Epidemiol. 2019 Mar 4;11:207-216. doi: 10.2147/CLEP.S178003. eCollection 2019. PMID 30881137
- [Result] Philip T, Guglielmi C, Hagenbeek A, Somers R, Van der Lelie H, Bron D, Sonneveld P, Gisselbrecht C, Cahn JY, Harousseau JL, et al. Autologous bone marrow transplantation as compared with salvage chemotherapy in relapses of chemotherapy-sensitive non-Hodgkin's lymphoma. N Engl J Med. 1995 Dec 7;333(23):1540-5. doi: 10.1056/NEJM199512073332305. PMID 7477169
- [Result] Gisselbrecht C, Glass B, Mounier N, Singh Gill D, Linch DC, Trneny M, Bosly A, Ketterer N, Shpilberg O, Hagberg H, Ma D, Briere J, Moskowitz CH, Schmitz N. Salvage regimens with autologous transplantation for relapsed large B-cell lymphoma in the rituximab era. J Clin Oncol. 2010 Sep 20;28(27):4184-90. doi: 10.1200/JCO.2010.28.1618. Epub 2010 Jul 26. PMID 20660832
- [Result] Mounier N, El Gnaoui T, Tilly H, Canioni D, Sebban C, Casasnovas RO, Delarue R, Sonet A, Beaussart P, Petrella T, Castaigne S, Bologna S, Salles G, Rahmouni A, Gaulard P, Haioun C. Rituximab plus gemcitabine and oxaliplatin in patients with refractory/relapsed diffuse large B-cell lymphoma who are not candidates for high-dose therapy. A phase II Lymphoma Study Association trial. Haematologica. 2013 Nov;98(11):1726-31. doi: 10.3324/haematol.2013.090597. Epub 2013 Jun 10. PMID 23753028
- [Result] Corazzelli G, Capobianco G, Arcamone M, Ballerini PF, Iannitto E, Russo F, Frigeri F, Becchimanzi C, Marcacci G, De Chiara A, Pinto A. Long-term results of gemcitabine plus oxaliplatin with and without rituximab as salvage treatment for transplant-ineligible patients with refractory/relapsing B-cell lymphoma. Cancer Chemother Pharmacol. 2009 Oct;64(5):907-16. doi: 10.1007/s00280-009-0941-9. Epub 2009 Feb 15. PMID 19219604
- [Result] Cazelles C, Belhadj K, Vellemans H, Camus V, Poullot E, Gaulard P, Veresezan L, Itti E, Becker S, Carvalho M, Dupuis J, Le Bras F, Lemonnier F, Roulin L, El Gnaoui T, Jardin F, Mounier N, Tilly H, Haioun C. Rituximab plus gemcitabine and oxaliplatin (R-GemOx) in refractory/relapsed diffuse large B-cell lymphoma: a real-life study in patients ineligible for autologous stem-cell transplantation. Leuk Lymphoma. 2021 Sep;62(9):2161-2168. doi: 10.1080/10428194.2021.1901090. Epub 2021 Mar 25. PMID 33764240
- [Result] Azizian NG, Li Y. XPO1-dependent nuclear export as a target for cancer therapy. J Hematol Oncol. 2020 Jun 1;13(1):61. doi: 10.1186/s13045-020-00903-4. PMID 32487143
- [Result] Gandhi UH, Senapedis W, Baloglu E, Unger TJ, Chari A, Vogl D, Cornell RF. Clinical Implications of Targeting XPO1-mediated Nuclear Export in Multiple Myeloma. Clin Lymphoma Myeloma Leuk. 2018 May;18(5):335-345. doi: 10.1016/j.clml.2018.03.003. Epub 2018 Mar 14. PMID 29610030
- [Result] Deng M, Zhang M, Xu-Monette ZY, Pham LV, Tzankov A, Visco C, Fang X, Bhagat G, Zhu F, Dybkaer K, Chiu A, Tam W, Zu Y, Hsi ED, Choi WWL, Huh J, Ponzoni M, Ferreri AJM, Moller MB, Parsons BM, van Krieken JH, Piris MA, Winter JN, Hagemeister F, Alinari L, Li Y, Andreeff M, Xu B, Young KH. XPO1 expression worsens the prognosis of unfavorable DLBCL that can be effectively targeted by selinexor in the absence of mutant p53. J Hematol Oncol. 2020 Nov 4;13(1):148. doi: 10.1186/s13045-020-00982-3. PMID 33148342
- [Result] Kalakonda N, Maerevoet M, Cavallo F, Follows G, Goy A, Vermaat JSP, Casasnovas O, Hamad N, Zijlstra JM, Bakhshi S, Bouabdallah R, Choquet S, Gurion R, Hill B, Jaeger U, Sancho JM, Schuster M, Thieblemont C, De la Cruz F, Egyed M, Mishra S, Offner F, Vassilakopoulos TP, Warzocha K, McCarthy D, Ma X, Corona K, Saint-Martin JR, Chang H, Landesman Y, Joshi A, Wang H, Shah J, Shacham S, Kauffman M, Van Den Neste E, Canales MA. Selinexor in patients with relapsed or refractory diffuse large B-cell lymphoma (SADAL): a single-arm, multinational, multicentre, open-label, phase 2 trial. Lancet Haematol. 2020 Jul;7(7):e511-e522. doi: 10.1016/S2352-3026(20)30120-4. PMID 32589977
- [Result] Kazim S, Malafa MP, Coppola D, Husain K, Zibadi S, Kashyap T, Crochiere M, Landesman Y, Rashal T, Sullivan DM, Mahipal A. Selective Nuclear Export Inhibitor KPT-330 Enhances the Antitumor Activity of Gemcitabine in Human Pancreatic Cancer. Mol Cancer Ther. 2015 Jul;14(7):1570-81. doi: 10.1158/1535-7163.MCT-15-0104. Epub 2015 May 1. PMID 25934708
- [Result] Corno C, Stucchi S, De Cesare M, Carenini N, Stamatakos S, Ciusani E, Minoli L, Scanziani E, Argueta C, Landesman Y, Zaffaroni N, Gatti L, Perego P. FoxO-1 contributes to the efficacy of the combination of the XPO1 inhibitor selinexor and cisplatin in ovarian carcinoma preclinical models. Biochem Pharmacol. 2018 Jan;147:93-103. doi: 10.1016/j.bcp.2017.11.009. Epub 2017 Nov 16. PMID 29155058
- See also: Related Info — http://ashpublications.org/blood/article/136/Supplement%201/11/471859/Selinexor-in-Combination-with-R-CHOP-for-Frontline
- See also: Related Info — http://www.semanticscholar.org/paper/Hitting-a-moving-target%3A-inhibition-of-the-nuclear-Sendino-Omaetxebarria/e3eebd3e1f9632d8cc3d012346a7f93dfc3bc906